CLINICAL TRIAL: NCT01006499
Title: Phase 4 Study of Role of 'Pentoxifylline and or IgM Enriched Intravenous Immunoglobulin in the Treatment of Neonatal Sepsis'
Brief Title: Role of 'Pentoxifylline and or IgM Enriched Intravenous Immunoglobulin in the Treatment of Neonatal Sepsis'
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Arzu Akdağ, ZTB
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-akdag
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Sepsis of the Newborn
Keywords: neonatal sepsis; pentoxyfilline; pentaglobin; biomarker; To reduce mortality in neonatal sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Pentoxifylline; pentaglobulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo group (Placebo Comparator): Receiving standard treatment plus placebo (5 mls/Kg of normal saline intravenously given over 4 hours).
  Interventions: Drug: Pentoxifylline, pentaglobin
- Pentoxifylline group (Active Comparator): Standard treatment plus 6 mg/Kg of Pentoxifylline intravenously (given over 4 hours) daily for three days.
  Interventions: Drug: Pentoxifylline, pentaglobin
- Pentaglobin group (Active Comparator): Standard treatment plus 250 mg/Kg of Pentaglobin intravenously (given over 4 hours) daily for three days
  Interventions: Drug: Pentoxifylline, pentaglobin
- Pentoxifylline plus Pentaglobin group (Active Comparator): Standard treatment plus 6 mg/Kg of Pentoxifylline plus 250 mg/Kg of Pentaglobin intravenously (given over 4 hours) daily for three days.
  Interventions: Drug: Pentoxifylline, pentaglobin

INTERVENTIONS:
Drug: Pentoxifylline, pentaglobin — Pentaglobin 250mg/kg/d over 4 hour for three days Pentoxyfilline 6mg/kg/h over 4 hour for three days Pentaglobin 250mg/kg/d over 4 hour for three days+Pentoxyfilline 6mg/kg/h over 4 hour for three days Placebo (normal saline 5ml/kg over 4 hour for three days

SUMMARY:
The investigators aim is to investigate whether adjuvant Pentoxifylline , IgM enriched IVIG or Pentoxifylline plus IgM-enriched IVIG reduced mortality from Neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria::

* All infants thought/diagnosed to have late or early onset sepsis.

Exclusion Criteria:

* Pentoxifylline or Pentaglobin has already been given
* Pentoxifylline or Pentaglobin is thought to be needed or contra-indicated
* Major congenital anomaly
* Intraventricular hemorrhage (Grade 3 veya 4)
* Congenital infections
* Inborn errors of metabolism

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
patient characteristics all cause mortality | two years
  Does adjuvant Pentoxifylline or Pentoxifylline plus IgM-enriched IVIG reduce mortality from Neonatal sepsis

SECONDARY OUTCOMES:
Neurodevelopmental morbidity secondary to sepsis at the age of 18 months Difference in biomarker levels | two years
  Assess the effectiveness of Pentoxifylline or Pentoxifylline plus IgM enriched IVIG in reducing neuro-developmental morbidity secondary to sepsis at the age of 18 months
Effect the production of pro-inflammatory bio-markers. | two years
  Whether Pentoxifylline or Pentoxifylline plus IgM enriched IVIG reduces the production of pro-inflammatory bio-markers

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak, Ankara, Turkey (Türkiye)